CLINICAL TRIAL: NCT00926380
Title: The Denosumab And Teriparatide Administration Study (DATA)
Brief Title: Denosumab, Teriparatide or Both for the Treatment of Postmenopausal Osteoporosis
Acronym: DATA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Benjamin Leder, MD, Principal Investigator, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20080723; 2009P000525
Record Dates: First submitted 2009-06-19; First posted 2009-06-23 (Estimated); Results first posted 2018-05-08 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-05

CONDITIONS: Osteoporosis
Keywords: osteoporosis; postmenopausal; denosumab; teriparatide; Forteo®; DXA; Bone Mineral Density; pQCT
MeSH Terms: conditions — Osteoporosis | interventions — Denosumab; Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- denosumab ONLY (Experimental)
  Interventions: Drug: denosumab
- teriparatide (Forteo®) ONLY (Experimental)
  Interventions: Drug: teriparatide
- denosumab and teriparatide (Forteo®) (Experimental)
  Interventions: Drug: denosumab; Drug: teriparatide

INTERVENTIONS:
Drug: denosumab — denosumab: 60 mg SC every 6 months
  Arms: denosumab ONLY; denosumab and teriparatide (Forteo®)
Drug: teriparatide — teriparatide: 20 mcg SC QD
  Other Names: Forteo®
  Arms: denosumab and teriparatide (Forteo®); teriparatide (Forteo®) ONLY

SUMMARY:
The aim of this study is to determine whether denosumab (an FDA-approved osteoporosis therapy), in combination with teriparatide (an FDA-approved osteoporosis therapy), will increase bone mineral density more than either one alone in postmenopausal osteoporotic women.

ELIGIBILITY:
Inclusion Criteria:

Must satisfy A and B and C and D below:

* (A) Women aged > 55
* (B) Postmenopausal
* (C) Osteoporotic with high risk of fracture

Exclusion Criteria:

* Confirmed serum alkaline phosphatase above upper normal limit with no explanation
* Liver disease (AST or ALT > 2 x upper normal limit).
* Renal disease (serum creatinine > 2.0 mg/dl).
* Hypercalcemia (Ca >10.5 mg/dL)
* Elevated blood PTH (intact PTH > 65 pg/ml)
* Serum 25-OH vitamin D < 20 ng/ml
* HCT < 32%.
* History of malignancy (except basal cell carcinoma) or radiation therapy.
* Significant cardiopulmonary disease including unstable coronary artery disease, stage D ACC/AHA heart failure or any other condition that the investigator deems may preclude the subject from participating safely or completing the protocol procedures.
* Major psychiatric disease that in the opinion of the investigator would preclude the subject from providing adequate informed consent or completing the protocol procedures.
* Excessive alcohol use or substance abuse that in the opinion of the investigator would preclude the subject from providing adequate informed consent or completing the protocol procedures.
* Known congenital or acquired bone disease other than osteoporosis (including osteomalacia, hyperparathyroidism, Paget's disease)
* Current use or use in the past 6 months of oral bisphosphonate
* Current use or use within the past 3 months of estrogens, selective estrogen receptor modulators, or calcitonin.
* Use of oral or parenteral glucocorticoids for more than 14 days within the past 6 months.
* Any current or previous use of strontium or any parenteral bisphosphonate.
* Known sensitivity to mammalian cell-derived drug products.
* Known sensitivity to teriparatide or any of its excipients.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2009-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Z Leder, MD, Principal Investigator — Massachusetts General Hospital; Robert M Neer, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Neer RM, Arnaud CD, Zanchetta JR, Prince R, Gaich GA, Reginster JY, Hodsman AB, Eriksen EF, Ish-Shalom S, Genant HK, Wang O, Mitlak BH. Effect of parathyroid hormone (1-34) on fractures and bone mineral density in postmenopausal women with osteoporosis. N Engl J Med. 2001 May 10;344(19):1434-41. doi: 10.1056/NEJM200105103441904. PMID 11346808
- [Background] Black DM, Greenspan SL, Ensrud KE, Palermo L, McGowan JA, Lang TF, Garnero P, Bouxsein ML, Bilezikian JP, Rosen CJ; PaTH Study Investigators. The effects of parathyroid hormone and alendronate alone or in combination in postmenopausal osteoporosis. N Engl J Med. 2003 Sep 25;349(13):1207-15. doi: 10.1056/NEJMoa031975. Epub 2003 Sep 20. PMID 14500804
- [Background] Finkelstein JS, Hayes A, Hunzelman JL, Wyland JJ, Lee H, Neer RM. The effects of parathyroid hormone, alendronate, or both in men with osteoporosis. N Engl J Med. 2003 Sep 25;349(13):1216-26. doi: 10.1056/NEJMoa035725. Epub 2003 Sep 20. PMID 14500805
- [Background] Cosman F, Nieves J, Woelfert L, Formica C, Gordon S, Shen V, Lindsay R. Parathyroid hormone added to established hormone therapy: effects on vertebral fracture and maintenance of bone mass after parathyroid hormone withdrawal. J Bone Miner Res. 2001 May;16(5):925-31. doi: 10.1359/jbmr.2001.16.5.925. PMID 11341338
- [Background] Kostenuik PJ, Capparelli C, Morony S, Adamu S, Shimamoto G, Shen V, Lacey DL, Dunstan CR. OPG and PTH-(1-34) have additive effects on bone density and mechanical strength in osteopenic ovariectomized rats. Endocrinology. 2001 Oct;142(10):4295-304. doi: 10.1210/endo.142.10.8437. PMID 11564687
- [Background] Lacey DL, Timms E, Tan HL, Kelley MJ, Dunstan CR, Burgess T, Elliott R, Colombero A, Elliott G, Scully S, Hsu H, Sullivan J, Hawkins N, Davy E, Capparelli C, Eli A, Qian YX, Kaufman S, Sarosi I, Shalhoub V, Senaldi G, Guo J, Delaney J, Boyle WJ. Osteoprotegerin ligand is a cytokine that regulates osteoclast differentiation and activation. Cell. 1998 Apr 17;93(2):165-76. doi: 10.1016/s0092-8674(00)81569-x. PMID 9568710
- [Background] Yasuda H, Shima N, Nakagawa N, Yamaguchi K, Kinosaki M, Mochizuki S, Tomoyasu A, Yano K, Goto M, Murakami A, Tsuda E, Morinaga T, Higashio K, Udagawa N, Takahashi N, Suda T. Osteoclast differentiation factor is a ligand for osteoprotegerin/osteoclastogenesis-inhibitory factor and is identical to TRANCE/RANKL. Proc Natl Acad Sci U S A. 1998 Mar 31;95(7):3597-602. doi: 10.1073/pnas.95.7.3597. PMID 9520411
- [Background] Bone HG, Bolognese MA, Yuen CK, Kendler DL, Wang H, Liu Y, San Martin J. Effects of denosumab on bone mineral density and bone turnover in postmenopausal women. J Clin Endocrinol Metab. 2008 Jun;93(6):2149-57. doi: 10.1210/jc.2007-2814. Epub 2008 Apr 1. PMID 18381571
- [Background] Miller PD, Bolognese MA, Lewiecki EM, McClung MR, Ding B, Austin M, Liu Y, San Martin J. Effect of denosumab on bone density and turnover in postmenopausal women with low bone mass after long-term continued, discontinued, and restarting of therapy: a randomized blinded phase 2 clinical trial. Bone. 2008 Aug;43(2):222-229. doi: 10.1016/j.bone.2008.04.007. Epub 2008 Apr 26. PMID 18539106
- [Background] Antoniucci DM, Sellmeyer DE, Bilezikian JP, Palermo L, Ensrud KE, Greenspan SL, Black DM. Elevations in serum and urinary calcium with parathyroid hormone (1-84) with and without alendronate for osteoporosis. J Clin Endocrinol Metab. 2007 Mar;92(3):942-7. doi: 10.1210/jc.2006-1788. Epub 2006 Dec 12. PMID 17164314
- [Derived] Tsai JN, Uihlein AV, Burnett-Bowie SM, Neer RM, Derrico NP, Lee H, Bouxsein ML, Leder BZ. Effects of Two Years of Teriparatide, Denosumab, or Both on Bone Microarchitecture and Strength (DATA-HRpQCT study). J Clin Endocrinol Metab. 2016 May;101(5):2023-30. doi: 10.1210/jc.2016-1160. Epub 2016 Mar 10. PMID 26964731
- [Derived] Leder BZ, Tsai JN, Uihlein AV, Wallace PM, Lee H, Neer RM, Burnett-Bowie SA. Denosumab and teriparatide transitions in postmenopausal osteoporosis (the DATA-Switch study): extension of a randomised controlled trial. Lancet. 2015 Sep 19;386(9999):1147-55. doi: 10.1016/S0140-6736(15)61120-5. Epub 2015 Jul 2. PMID 26144908
- [Derived] Yu EW, Kumbhani R, Siwila-Sackman E, DeLelys M, Preffer FI, Leder BZ, Wu JY. Teriparatide (PTH 1-34) treatment increases peripheral hematopoietic stem cells in postmenopausal women. J Bone Miner Res. 2014 Jun;29(6):1380-6. doi: 10.1002/jbmr.2171. PMID 24420643
- [Derived] Tsai JN, Uihlein AV, Lee H, Kumbhani R, Siwila-Sackman E, McKay EA, Burnett-Bowie SA, Neer RM, Leder BZ. Teriparatide and denosumab, alone or combined, in women with postmenopausal osteoporosis: the DATA study randomised trial. Lancet. 2013 Jul 6;382(9886):50-6. doi: 10.1016/S0140-6736(13)60856-9. Epub 2013 May 15. PMID 23683600

RESULTS

PARTICIPANT FLOW:
Period: Year 1
Arm/Group | Denosumab ONLY | Teriparatide (Forteo®) ONLY | Denosumab and Teriparatide (Forteo®)
Started | 33 | 31 | 30
Completed | 33 | 30 | 29
Not Completed | 0 | 1 | 1
Period: Year 2
Arm/Group | Denosumab ONLY | Teriparatide (Forteo®) ONLY | Denosumab and Teriparatide (Forteo®)
Started | 33 | 30 | 29
Completed | 31 | 28 | 24
Not Completed | 2 | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Denosumab ONLY | Teriparatide (Forteo®) ONLY | Denosumab and Teriparatide (Forteo®) | Total
Number analyzed (Participants) | 33 | 31 | 30 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (8.3) | 65.5 (7.9) | 65.9 (9.0) | 65.9 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 31 | 30 | 94
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 32 | 31 | 29 | 92
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 3
  White | 31 | 31 | 28 | 90
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 31 | 30 | 94
Body-mass index [Mean (Standard Deviation); unit: kg/m^2] | 24.1 (3.9) | 25.5 (3.8) | 25.4 (4.9) | 25.0 (4.2)
History of fragility fracture [Count of Participants; unit: Participants] | 12 | 16 | 10 | 38
Previous oral bisphosphonate use [Count of Participants; unit: Participants] | 12 | 13 | 10 | 35
25-Hydroxyvitamin D (ng/mL) [Mean (Standard Deviation); unit: ng/mL] | 35.3 (10.5) | 31.2 (8.5) | 33.9 (11.8) | 33.5 (10.5)
Alkaline phosphatase concentration in serum (U/L) [Mean (Standard Deviation); unit: U/L] | 78.8 (16.8) | 75.8 (16.8) | 84.2 (20.8) | 79.6 (18.4)
Osteocalcin (ng/mL) [Mean (Standard Deviation); unit: ng/mL] | 42.9 (19.4) | 49.0 (28.8) | 52.2 (29.9) | 47.8 (26.2)
Serum amino-terminal propeptide of type 1 procollagen (P1NP) (µg/L) [Mean (Standard Deviation); unit: µg/L] | 45.7 (16.7) | 46.0 (19.5) | 49.3 (20.9) | 47.1 (19.0)
Serum β-C-terminal telopeptide of type 1 collagen (CTX) (ng/mL) [Mean (Standard Deviation); unit: ng/mL] | 0.39 (0.21) | 0.36 (0.15) | 0.43 (0.17) | 0.39 (0.18)
DXA Bone Density (g/cm^2) (Posterior-anterior lumbar spine) [Mean (Standard Deviation); unit: g/cm^2] | 0.866 (0.088) | 0.823 (0.111) | 0.856 (0.131) | 0.848 (0.112)
DXA Bone Density (g/cm^2) (Femoral neck) [Mean (Standard Deviation); unit: g/cm^2] | 0.641 (0.086) | 0.643 (0.061) | 0.642 (0.067) | 0.642 (0.071)
DXA Bone Density (g/cm^2) (Total hip) [Mean (Standard Deviation); unit: g/cm^2] | 0.766 (0.100) | 0.757 (0.068) | 0.759 (0.073) | 0.761 (0.081)
DXA Bone Density (g/cm^2) (Distal 1/3 of the radius shaft) [Mean (Standard Deviation); unit: g/cm^2] | 0.602 (0.082) | 0.612 (0.069) | 0.613 (0.070) | 0.609 (0.073)

OUTCOME MEASURES:

1. Primary Outcome: Change in Spine Bone Density From Baseline to 2 Years
Time Frame: Baseline and 2 years
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Denosumab ONLY | Teriparatide (Forteo®) ONLY | Denosumab and Teriparatide (Forteo®)
Number analyzed (Participants) | 33 | 31 | 30
percent change | 8.3 (3.4) | 9.5 (5.9) | 12.9 (5.0)

ADVERSE EVENTS:
Arm/Group | Denosumab ONLY | Teriparatide (Forteo®) ONLY | Denosumab and Teriparatide (Forteo®)
Serious Adverse Events (participants affected / at risk) | 1/33 | 2/31 | 1/30
Other Adverse Events (participants affected / at risk) | 4/33 | 5/31 | 4/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab ONLY (N=33) | Teriparatide (Forteo®) ONLY (N=31) | Denosumab and Teriparatide (Forteo®) (N=30)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Heart attack (Cardiac disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab ONLY (N=33) | Teriparatide (Forteo®) ONLY (N=31) | Denosumab and Teriparatide (Forteo®) (N=30)
Rash (Skin and subcutaneous tissue disorders) | 4 | 0 | 2
Reactions at injection site (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Hypercalcemia (Endocrine disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No